CLINICAL TRIAL: NCT04932369
Title: The Effect of Emotion Regulation Training on Anxiety, in College Students in Egypt During COVID-19
Brief Title: The Effect of Emotion Regulation Training on Anxiety, in College Students in Egypt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, Amani Safwat Albrazi, Dr, British University In Egypt
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CL-2008
Record Dates: First submitted 2021-06-12; First posted 2021-06-21 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Anxiety; Emotion Regulation
Keywords: University's students; COVID-19
MeSH Terms: conditions — Anxiety Disorders; Emotional Regulation; COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ER GROUP (Experimental): The training sessions were based on the Dialectical Behavior Therapy Skills (Linehan, 2015). Each group received eight 90-min sessions of the emotion regulation training (one session per week) carried out by qualified clinical psychologist. The training includes group gathering, homework and telephone consultation as needed.
  Interventions: Behavioral: Emotion Regulation training based on DBT
- Control group (No Intervention): They completed two assessments, 3-months apart

INTERVENTIONS:
Behavioral: Emotion Regulation training based on DBT — trained about emotion regulation and problem solving during eight 90-min group sessions
  Arms: ER GROUP

SUMMARY:
The important role of Emotion Regulation (ER) in managing stress and anxiety is well recognized. Aims: 1) assessing the level of anxiety, and the level of difficulties in emotion regulation (DER) among University Students during COVID-19, 2) investigating the effect of the emotional regulation training program on the anxiety of University Students during the COVID-19. Methods: Part I, students will be assessed for their anxiety, DER, and the general impact of COVID-19 on their lives. The students will complete Beck Anxiety Inventory (BAI) and Difficulties in Emotion Regulation Scale (DERS). Part II will be a Randomized Control Trial (RCT) using a pre-assessment and a post-assessment. A voluntary sample of students will randomly assigned to either a group that will receive emotion regulation training or a control group. The training program is an adapted version of DBT skills training. The training program will include mindfulness, emotion regulation, and problem-solving skills through eight 90- min group sessions.

ELIGIBILITY:
Inclusion Criteria:

* Being an active student at the University

Exclusion Criteria:

1. Receiving treatment at the hospital during the time that the study was in progress
2. Having been diagnosed with psychotic disorders
3. Having mental retardation

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Change in anxiety from Baseline to the completion of training three months later using Beck Anxiety Inventory (BAI) | 3 months. Assessments of anxiety will be collected from all students two times, three months apart
  Beck Anxiety Inventory (BAI): was developed by Dr. Aaron T. Beck and it is a brief measure of anxiety with a focus on somatic symptoms of anxiety such as nervousness, dizziness, inability to relax (Beck et al., 1988). It has a total of 21 items that takes approximately 10-15 minutes to complete. Answers are on a 4-point Likert scale and range from 0 (not at all) to 3 (severely). The values for each item are added together to get an overall or total score for all 21 symptoms that can vary from 0 to 63 points. A total score of 0 - 7 indicates "Minimal" anxiety; 8 - 15 indicates "Mild" anxiety; 16 -25 indicates "Moderate" anxiety; and 26 - 63 indicates "Severe" anxiety
Change in difficulties in emotion regulation from Baseline to the completion of training three months later using Emotion regulation difficulties Scale | 3 months. Assessments of DER will be collected from all students two times, three months apart
  The DERS is a 36-item self-reported questionnaire that assesses an individual's ability to regulate their emotions (Gratz & Roemer, 2004). Participants rate items on a 5-point Likert scale (1 = seldom to 5 = nearly frequently) to represent their self-perceived reactions to stressful emotional situations. The DERS produces an overall difficulty score in ER as well as six subscales: (a) Awareness, (b) Clarity, (c) Nonacceptance, (d) Impulsivity, (e) Goals, and (f) Strategies. Subscales are evaluated in such a way that higher values imply more difficulty.

CONTACTS AND LOCATIONS:
Overall Officials: Amani Elbarazi, Ph.D., Principal Investigator — The British University in Egypt
Locations (1):
- The British university in Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No